CLINICAL TRIAL: NCT05944822
Title: Study of Pro-inflammatory Cytokines in Case of Essure® Contraceptive Implants
Brief Title: Pro-inflammatory Cytokines in Case of Essure®
Acronym: ESCYTO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0557
Record Dates: First submitted 2023-06-27; First posted 2023-07-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-07

CONDITIONS: Inflammatory Disease
Keywords: contraceptive implants; pro-inflammatory cytokines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Essure: patient who underwent removal of the Essure® contraceptive implant
  Interventions: Other: pro-inflammatory cytokines
- Control with no endometriosis/adenomyosis: patient who underwent benign laparoscopic gynecological surgery and with no diagnosis of endometriosis or adenomyosis
  Interventions: Other: pro-inflammatory cytokines
- Control with endometriosis/adenomyosis: patient who underwent benign laparoscopic gynecological surgery and with diagnosis of endometriosis or adenomyosis
  Interventions: Other: pro-inflammatory cytokines

INTERVENTIONS:
Other: pro-inflammatory cytokines — compare the levels of pro-inflammatory cytokines in patients with Essure® contraceptive implants and in control patients with endometriosis or adenomyosis.

SUMMARY:
It is estimated that 750,000 women (including 200,000 French) have benefited from permanent sterilization by ESSURE® contraceptive implant. The observation in some of these patients of gynecological and extra-gynecological symptoms leads to the surgical removal of these implants.

The pathophysiological mechanism(s) is (are) not yet determined. Several pathophysiological hypotheses have been proposed, in particular the inflammatory hypothesis. The investigators propose to study markers of inflammation (pro-inflammatory cytokines) in peritoneal fluid and blood. Cytokines are involved in the physiopathology of autoimmune diseases, infectious pathologies, or even cancer; they are used in everyday practice and can constitute a therapeutic target.

Based on the literature which finds a high concentration of cytokines in cases of endometriosis, and a low concentration in healthy control patients, the investigators want to assess inflammation in patients with Essure® implants.

The demonstration of one or more specifically increased cytokines in the Essure® group could validate the inflammatory hypothesis and lead to the implementation of specific treatments and relevant markers.

ELIGIBILITY:
Inclusion Criteria:

* women over 18
* intervention between January 2021 and November 2022
* person having expressed his non-opposition

Essure group : patient who underwent removal of the Essure® contraceptive implant

Control with no endometriosis/adenomyosis : patient who underwent benign laparoscopic gynecological surgery and with no diagnosis of endometriosis or adenomyosis

Control with endometriosis/adenomyosis : patient who underwent benign laparoscopic gynecological surgery and with diagnosis of endometriosis or adenomyosis

Exclusion Criteria:

* inability to understand the information given
* person deprived of liberty
* person under guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This study focuses on patients who underwent surgery to remove the Essure® contraceptive implant and on control patients who underwent benign gynecological laparoscopic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
cytokine IL10 in peritoneal fluid | through study completion, an average of 4 months
  Level of cytokine IL10 in peritoneal fluid

CONTACTS AND LOCATIONS:
Locations (1):
- Gynaecology Department, Hôpital Femme Mère Enfant Hospices Civisl de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No